CLINICAL TRIAL: NCT00044954
Title: Low Dose Total-Body Irradiation And Fludarabine Followed By HLA Matched Allogeneic Stem Cell Transplantation For Hematologic Malgnancies - A Multi-Center Study
Brief Title: Total-Body Irradiation, Fludarabine, and Peripheral Stem Cell Transplantation in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069461; UTSMC-0799296; AMGEN-UTSMC-0799296; IBMTR-SC-00-03.1; ROCHE-UTSMC-0799296; SPRI-UTSMC-0799296; NCI-V02-1705
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: recurrent adult Hodgkin lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; adult acute myeloid leukemia in remission; recurrent grade 3 follicular lymphoma; recurrent adult diffuse large cell lymphoma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; recurrent mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; refractory multiple myeloma; stage I mantle cell lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; refractory chronic lymphocytic leukemia; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Hodgkin Disease; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Leukemia, Lymphocytic, Chronic, B-Cell; Congenital Abnormalities | interventions — Cyclosporine; fludarabine phosphate; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: therapeutic allogeneic lymphocytes
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: mycophenolate mofetil
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage cancer cells. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with donor peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining total-body irradiation with fludarabine and donor peripheral stem cell transplantation in treating patients who have hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate and duration of response in patients with low-risk hematologic malignancies treated with low-dose total-body irradiation (TBI) and fludarabine followed by HLA-matched allogeneic stem cell transplantation followed by a slow immunosuppression taper and donor leukocyte infusions (DLI).
* Determine the response rate and duration of response in patients with high-risk hematologic malignancies treated with low-dose TBI and fludarabine followed by HLA-matched allogeneic stem cell transplantation followed by a faster immunosuppression taper and DLI.
* Determine the incidence and extent of graft-versus-host disease, regimen-related toxicity, and engraftment in patients treated with these regimens.
* Assess the quality of life of patients treated with these regimens.

OUTLINE: This is a multicenter study. Patients are assigned to 1 of 2 groups (high-risk vs low-risk hematologic malignancy). The high-risk group includes acute myelogenous leukemia, myelodysplastic syndromes, accelerated phase chronic myelogenous leukemia (CML), second chronic phase CML, and non-Hodgkin's lymphoma. The low-risk group includes Hodgkin's lymphoma, first chronic phase CML, multiple myeloma, and chronic lymphocytic leukemia.

Patients receive fludarabine IV on days -4 to -2. Patients undergo total-body irradiation on day 0 followed by allogeneic stem cell transplantation. Patients also receive oral mycophenolate mofetil on days 0-28.

High-risk patients receive oral cyclosporine twice daily on days -2 to day 60. Patients with persistent disease, T-cell chimerism, and no graft-vs-host disease (GVHD) on day 90 receive up to 3 doses of donor leukocyte infusion (DLI) over the next 4 months.

Low-risk patients receive oral cyclosporine twice daily on days -2 to day 150. Patients with persistent disease, T-cell chimerism, and no GVHD on day 180 receive up to 3 doses of DLI over the next 4 months.

Quality of life is assessed at baseline and at 1, 3, 6, 9, 12, 18, and 24 months.

Patients are followed at 1, 3, 6, 9, and 12 months and then annually for 2 years.

PROJECTED ACCRUAL: A total of 120 patients (60 per group) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following hematologic malignancies:

  * Chronic myelogenous leukemia (CML)

    * First or second chronic phase
    * Accelerated phase
  * Acute myelogenous leukemia (AML)

    * At least second remission
    * First remission allowed if poor-risk features are present (complex chromosome karyotype, abnormalities of chromosomes, especially 5 or 7, 12p-, +13, +8, t[9:11])
  * Myelodysplastic syndromes (MDS)

    * Intermediate- or high-risk disease by the prognostic scoring system
  * Multiple myeloma (MM)
  * Hodgkin's lymphoma

    * Second or greater relapse
    * First relapse allowed if disease-free interval is less than 1 year
    * Ineligible for autologous transplantation
  * Non-Hodgkin's lymphoma (NHL)

    * Grade III follicular large cell (relapsed after one course of prior chemotherapy)
    * Diffuse large cell (relapsed after one course of prior chemotherapy)
    * Mantle cell
  * Chronic lymphocytic leukemia (CLL)

    * Relapsed after at least 1 course of prior therapy
* Must have 6 out of 6 HLA A-, B-, and DR- identical sibling donor

PATIENT CHARACTERISTICS:

Age

* 18 to 75 for patients with MM
* 50 to 75 for patients with CML, AML, MDS, Hodgkin's lymphoma, NHL, or CLL
* 18 to 49 for patients with CML, AML, MDS, Hodgkin's lymphoma, NHL, or CLL who are considered eligible for an allogeneic bone marrow transplantation (BMT) but do not meet institutional criteria for a standard allogeneic BMT

Performance status

* Zubrod 0-2

Life expectancy

* At least 6 months

Hematopoietic

* Not specified

Hepatic

* Bilirubin no greater than 3 mg/dL

Renal

* Creatinine no greater than 2 mg/dL

Cardiovascular

* LVEF at least 40% by MUGA or echocardiogram

Pulmonary

* DLCO at least 50% of predicted

Other

* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No recent history of drug or alcohol abuse
* No other prior malignancy except basal cell skin cancer
* No uncontrolled bacterial, viral, fungal, or parasitic infections

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior autologous transplantation allowed if disease progression occurred
* No prior or concurrent tandem autologous transplantation followed by non-myeloablative-allograft protocol

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-11 (Actual); Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert H. Collins, MD, Study Chair — Simmons Cancer Center
Locations (14):
- United States (14):
  - Rocky Mountain Cancer Centers - Denver Midtown, Denver, Colorado
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Kansas City Cancer Centers - Central, Kansas City, Missouri
  - Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin